CLINICAL TRIAL: NCT06612320
Title: Refusal to Participate in a Randomized Trial Involving Pregnancy and Childbirth: Factors Associated with Refusal and Reasons for Refusal and Acceptance
Acronym: REFWIT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240778
Record Dates: First submitted 2024-09-06; First posted 2024-09-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy Related
Keywords: Refusal; clinical trial; factors; reasons; pregnancy; pre-eclampsia
MeSH Terms: conditions — Treatment Refusal; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acceptance: Women who accept to participate to a Randomized Controlled Trial (RCT)
  Interventions: Behavioral: Questionnaire about acceptance
- Refusal: Women who refuse to participate to a Randomized Controlled Trial (RCT)
  Interventions: Behavioral: Questionnaire about refusal

INTERVENTIONS:
Behavioral: Questionnaire about acceptance — Questionnaire about acceptance
  Groups: Acceptance
Behavioral: Questionnaire about refusal — Questionnaire about refusal
  Groups: Refusal

SUMMARY:
The main objective is to assess whether there are factors associated with women's refusal to participate in a randomized clinical trial involving pregnancy and childbirth in France. The secondary objective is to qualitatively evaluate the reasons for acceptance and refusal to participate.

DETAILED DESCRIPTION:
1. Determine the acceptance/refusal rate among all women identified, eligible and offered RCT.
2. Comparison of demographic characteristics between the two groups

   * Group 1: women accepting to participate in RCT
   * Group 2: women refusing to participate in RCT
3. Assessment of motivations for acceptance (based on questionnaire given to women who agree to participate)
4. Evaluation of reasons for refusal to participate - obstacles (based on the questionnaire given to women who refuse to participate).

ELIGIBILITY:
Inclusion Criteria:

The study will be offered to all women who have been offered to participate in a randomized trial relating to their pregnancy and/or childbirth in participating services.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to all women who have been offered to participate in a randomized trial relating to their pregnancy and/or childbirth in participating services.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Collection of maternal demographic characteristics | Day 1
  Age, level of education, profession, geographic origin, health insurance/mutual, marital status The primary objective is to assess whether there are factors associated with women's refusal to participate in randomized clinical trials.
  No score, it is a qualitative analyse.
Collection of obstetric characteristics | Day 1
  Parity, obstetric history (first-trimester pregnancy loss, IUFD, perinatal death), pregnancy complications, gestational age… The primary objective is to assess whether there are factors associated with women's refusal to participate in randomized clinical trials.
  No score, it is a qualitative analyse.
Collection of characteristics related to information provided | Day 1
  By whom? , with whom? (impact of the companion), when? The primary objective is to assess whether there are factors associated with women's refusal to participate in randomized clinical trials.
  No score, it is a qualitative analyse.

SECONDARY OUTCOMES:
Motivation linked to acceptance | Day 1
  Evaluation of motivation linked to acceptance (based on the questionnaire given to women who agree to participate).
  No score, it is a qualitative analyse.
Reason for refusing to participate | Day 1
  Evaluation of the reason for refusing to participate (based on the questionnaire given to women who refuse to participate)
  No score, it is a qualitative analyse.

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Athiel, MD, Principal Investigator — Port-Royal Maternity - APHP
Locations (4):
- France (4):
  - APHP - Antoine Béclère hospital - Maternity, Clamart, IDF
  - APHP - Louis Mourier hospital - Maternity, Colombes, IDF
  - APHP - Trousseau Hospital - Gynecology-Obstetrics-Maternity, Paris, IDF
  - APHP - Port-Royal Maternity, Paris, IDF

IPD SHARING:
Plan to Share IPD: No